CLINICAL TRIAL: NCT02234921
Title: A Pilot Study of DPV-001 DRibble Vaccine With Imiquimod in Advanced Prostate Cancer
Brief Title: Pilot Study of DRibble Vaccine for Prostate Cancer Patients
Acronym: DRibble
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UbiVac (Industry)
Collaborators: Providence Health & Services (Other); Providence Cancer Center (Unknown); Providence Cancer Center, Earle A. Chiles Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-116B
Record Dates: First submitted 2014-09-04; First posted 2014-09-09 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Adenocarcinoma of the Prostate
Keywords: Prostate; Adenocarcinoma; Metastatic; DRibble; Immunotherapy; Microbiome
MeSH Terms: conditions — Adenocarcinoma; Neoplasm Metastasis; Sialorrhea | interventions — Cyclophosphamide; Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DRibble Vaccine (Experimental): Patients will receive cyclophosphamide 3 days prior to the first of 9 planned DRibble vaccine injections. Imiquimod will be applied following 6 injections. Patients will receive 2 HPV vaccinations (Human papillomavirus).
  Interventions: Drug: Cyclophosphamide; Biological: DRibble Vaccine; Biological: HPV Vaccinations; Drug: Imiquimod

INTERVENTIONS:
Drug: Cyclophosphamide — A single dose of cyclophosphamide, 300 mg/m2, will be administered intravenously 3 Days prior to the first vaccine.
  Other Names: Cytoxan
Biological: DRibble Vaccine — DRibble vaccine will be administered at Weeks 1, 4, 7, 10, 13, 16, 19 and 22. Eight vaccinations will be administered. Week 1 and 4 vaccines will be administered by intranodal injections performed using ultrasound guidance.
  Other Names: DPV-001 DRibble vaccine
Biological: HPV Vaccinations — Patients will receive a dose of 0.5-mL CERVARIX at week 1 (Day 4) and week 7 by intramuscular injection at a site distant from the DRibble vaccine.
  Other Names: Ceravix
Drug: Imiquimod — Imiquimod cream (5%, 250 mg) will be self-applied topically for 5 consecutive days by patients to a 4 x 5-cm outlined area of healthy extremity skin starting on the day of the second vaccine and again during each additional vaccine cycle.

SUMMARY:
This is a pilot study of the DRibble vaccine in patients with advanced prostate cancer.

DETAILED DESCRIPTION:
The primary objective of this pilot study is to assess the safety and tolerability of DRibble vaccine, cyclophosphamide, imiquimod, and Ceravix in castrate resistant prostate cancer.

This study will also assess:

* the immune profile of tumor biopsy specimens if sites amenable to biopsy are present
* humoral and cellular responses to cancer antigens after DRibble vaccination
* the response to a reporter antigen vaccine (Ceravix) after DRibble vaccination

An exploratory objective is to characterize the microbiome before and after study drugs administration and correlate prostate cancer responses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have measurable or evaluable metastatic castrate resistant adenocarcinoma of the prostate with progression after chemotherapy, combined androgen blockade and/or peripheral androgen or androgen receptor suppression. Either histologic or serum marker diagnosis is acceptable.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Ability to give informed consent and comply with the protocol.
* Prior therapy with investigational agents must have been completed at least 3 weeks prior to study enrollment.
* Patients must have normal organ and marrow function as determined by routine blood tests

Exclusion Criteria:

* Active autoimmune disease except vitiligo or hypothyroidism.
* Active other malignancy.
* Known HIV positive and/or Hepatitis B or C positive.
* Other medical or psychiatric conditions that in the opinion of the Principal Investigator would preclude safe participation in protocol.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-10-24 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Safety Assessment | 28 Weeks
  Patients will come to clinic 10 times over a 28 week period and have blood tests and vital sign measurements at each visit. In addition, patients will have 8 physical exams and performance status evaluations during this time period to evaluate possible toxicities related to study treatment.

SECONDARY OUTCOMES:
Immune Response | 28 weeks
  Patients will have 11 blood draws during the study to evaluate the immune response. In addition, patients will undergo two leukapheresis procedures and provide two biopsy samples (if cancer is amenable to safe biopsy) to evaluate immune response.
Prostate Cancer Response to DRibble vaccine | 28 weeks
  Patients will have 8 Prostate-Specific Antigen (PSA) Tests over a 22-week period and 3 CT scans over a 28-week period to assess response to treatment.

OTHER OUTCOMES:
Microbiome identification | 12 weeks
  Patients will provide 3 stool samples for microbiome identification for future research to see if there is a correlation with response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Curti, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Health & Services, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Providence Cancer Center — http://oregon.providence.org/our-services/p/providence-cancer-center/